CLINICAL TRIAL: NCT06131736
Title: Comparative Effects of High Intensity Interval Training and Cluster Training on Speed, Explosive Strength and Functional Performance in Football Players.
Brief Title: Effects of High Intensity Interval Training and Cluster Training on Speed, Explosive Strength and Functional Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0431
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: High Intensity Interval Training; Functional Performance; Football Players
Keywords: Explosive Strength, High Intensity Interval Training, Speed

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The Assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tabata Training (Experimental): HIIT training programs follow Tabata protocol. This protocol was created with the aim of improving the aerobic and anaerobic characteristics beyond the threshold (anaerobic). It consists of performing seven or eight repetitions at maximum intensity, alternating with ten seconds of passive recovery. The series lasts approximately four minutes (240 sec). Given the intensity of the Tabata protocol, it is necessary to finish the workout with a cool down of at least 10-15 minutes. It includes exercises like push-ups, split squats, box jumps, burpees, jumping rope, jumping jacks and more. This training program, lasting about 20 minutes, was repeated three times a week for a total of 6 weeks. The duration of this type of work is not accidental. In fact, it has been scientifically established that only after this period it is possible to find significant improvements in speed, strength and functional activity
  Interventions: Other: Tabata Training
- Cluster Traning (Experimental): The cluster training consist squat, leg extension, leg curl, heel raise, French curl, barbell curl, Bench press, Incline bench press, behind the neck press with barbell, Overhead press with barbell. The movements were performed in 3 sets, each set containing 9 repetitions with 60-90 seconds of rest between each two sets. Each training session consisted of three steps: Warm up Basic training and Cool-down. Both groups performed the first and the third stage in 10 minutes
  Interventions: Other: Cluster Training

INTERVENTIONS:
Other: Tabata Training — This training program, lasting about 20 minutes, was repeated three times a week for a total of 6 weeks.
  Arms: Tabata Training
Other: Cluster Training — The movements were performed in 3 sets, each set containing 9 repetitions with 60-90 seconds of rest between each two sets.
  Arms: Cluster Traning

SUMMARY:
High-intensity interval training has been beneficial in many sports and significantly enhanced the results of physical training. Consequently, it has progressively been implemented among the football players. A Cluster Set (CS) is a set that has been broken up into smaller blocks of repeats with the inclusion of brief intra-set breaks or a reorganization of the breaks between repetitions. The initial assumption is that this design would offer a superior rise in exercise quality with the potential to maintain or enhance performance and enable larger loads, leading to stronger performance adaptations. The objective of the study is to compare the effects of high intensity interval training and cluster training on speed, explosive strength and functional performance in football players.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of high intensity interval training and cluster training on speed, explosive strength and functional performance in football players.This is randomized clinical trial that will be conducted at football club, Pakistan sport club Lahore. Non-Probability convenient sampling technique will be used to collect data. The study will be completed in 6 months after the approval of ethical committee of RCRS & Allied Health Sciences. Total number of participants will be 54, in group A participants will be 27, in group B participants will be 27. Performance, speed and strength will be measured by using FMS, 30-meter speed test and vertical jump test respectively. The participants will be divided into two groups. Group A will receive high intensity interval training (HIIT) and group B will receive cluster training. The training program will be conducted for 6 weeks and data will be collected pre and post training session. The data will be entered and analyzed using SPSS version 25 and Shapiro wilk test will be applied to determine the normality of the data. If data will be normally distributed then parametric type of statistical test will be applied while if the data will not normally distribute then non parametric type of test will be applied.

ELIGIBILITY:
Inclusion Criteria:

* • Male Players

  * Age between 18-30 years
  * At least 1 years of football experience

Exclusion Criteria:

* • Individuals with a lower extremity injury

  * Vestibular problems
  * Visual problems
  * Individuals who have had a concussion within the past 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
FMS (Functional movement screen) | Pre And 6 Weeks Post
  The FMS assesses seven fundamental movement patterns that require mobility and stability of the body and limb. These seven movements include the 1) Deep squat (DS) 2) Hurdle step (HS) 3) In-line lunge (IL) 4) Active straight leg raise (ASLR) 5) Trunk push-up (TP) 6) Rotary stability (RS) and 7) Shoulder mobility. Each movement in the FMS is rated by an assessor from 0 to 3 based on their ability to perform the movements without compensatory actions.
30 METER SPRINT TEST | Pre And 6 Weeks Post
  The purpose of this test is to determine acceleration, maximum running speed and speed endurance, depending on the distance run. The test involves running a single maximum sprint over 30 meters, with the time recorded.
THE VERTICAL JUMP TEST | Pre And 6 Weeks Post
  A vertical jump test gauge is used to conduct the test. Applicants should stand with their feet level and hip width apart beneath the testing gauge, with their dominant side closer to the gauge. The person then raises their dominant arm and fingers vertically over their head. On the test gauge, the test assessor then set the applicant's reach height to zero (0). The leap must be done with both feet flat on the ground without taking a step or running up from the starting position. To safeguard their lower limbs, candidates must take off and land with both feet. Only two (2) tries are permitted for applicants who must leap 30cm or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Arslan Sarwar, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- PSB-Coaching Centre, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sainani KL, Borg DN, Caldwell AR, Butson ML, Tenan MS, Vickers AJ, Vigotsky AD, Warmenhoven J, Nguyen R, Lohse KR, Knight EJ, Bargary N. Call to increase statistical collaboration in sports science, sport and exercise medicine and sports physiotherapy. Br J Sports Med. 2021 Jan;55(2):118-122. doi: 10.1136/bjsports-2020-102607. Epub 2020 Aug 19. No abstract available. PMID 32816788
- [Background] Thorborg K, Mendonca L. Sports Physiotherapy for All. Int J Sports Phys Ther. 2021 Oct 1;16(5):1178-1180. doi: 10.26603/001c.28268. eCollection 2021. No abstract available. PMID 34631240
- [Background] Arslan E, Orer GE, Clemente FM. Running-based high-intensity interval training vs. small-sided game training programs: effects on the physical performance, psychophysiological responses and technical skills in young soccer players. Biol Sport. 2020 Jun;37(2):165-173. doi: 10.5114/biolsport.2020.94237. Epub 2020 Mar 31. PMID 32508384
- [Background] Zaras N, Stasinaki AN, Mpampoulis T, Spiliopoulou P, Hadjicharalambous M, Terzis G. Effect of Inter-Repetition Rest Vs. Traditional Resistance Training on The Upper Body Strength Rate of Force Development and Triceps Brachii Muscle Architecture. J Hum Kinet. 2022 Feb 10;81:189-198. doi: 10.2478/hukin-2022-0016. eCollection 2022 Jan. PMID 35291627
- [Background] Kunz P, Engel FA, Holmberg HC, Sperlich B. A Meta-Comparison of the Effects of High-Intensity Interval Training to Those of Small-Sided Games and Other Training Protocols on Parameters Related to the Physiology and Performance of Youth Soccer Players. Sports Med Open. 2019 Feb 21;5(1):7. doi: 10.1186/s40798-019-0180-5. PMID 30790134
- [Background] Nickerson BS, Williams TD, Snarr RL, Park KS. Individual and Combined Effect of Inter-repetition Rest and Elastic Bands on Jumping Potentiation in Resistance-Trained Men. J Strength Cond Res. 2019 Aug;33(8):2087-2093. doi: 10.1519/JSC.0000000000002593. PMID 29863591